CLINICAL TRIAL: NCT06562257
Title: Honey as A Wound Care Modality in Treating Deep Neck Space Abscess: A Randomized Clinical Trial
Brief Title: Honey as A Wound Care Modality in Treating Deep Neck Space Abscess
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gadjah Mada University (Other)
Responsible Party: Principal Investigator, DIAN PARAMITA WULANDARI, Principal Investigator, Gadjah Mada University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KE/FK/0668/EC/2024
Record Dates: First submitted 2024-08-14; First posted 2024-08-20 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Neck Abscess
Keywords: Deep neck space infection; Deep neck space abscess; Wound healing; Honey dressing; Bates Jensen Wound Assessment Tool
MeSH Terms: interventions — Honey

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Both patients and the principal investigator will remain blinded throughout the completed treatment period. Treatment allocations will only be disclosed after the final database lock. The patients are primarily handled by a principal investigator and resident doctor who is in charge of the evaluation of inclusion or exclusion criteria, adverse events, relapses, and side effects
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Group (Standard Dressing and Honey) (Experimental): In the treatment group, we combined standard procedures with the application of Nusantara Honey. A 120 cm gauze roll was soaked in a bowl containing 12 cc of Nusantara Honey for precisely 1 minute until saturation. Once the wound bed had risen sufficiently, the honey-soaked gauze was applied and covered with sterile gauze.
  Interventions: Other: Honey; Other: PHMB Solution
- Control Group (Standard Dressing) (Active Comparator): The control group adhered to the established standard operating procedure (SOP) at the Larynx Pharynx subdivision of Dr. Sardjito Hospital. This protocol involved several steps of wound debridement, saline irrigation, gauze roll application, and Prontosan administration.
  Interventions: Other: PHMB Solution

INTERVENTIONS:
Other: Honey — Honey has a long-standing reputation for promoting wound healing and offers a more economical treatment modality. Nusantara Honey, a GMP-certified product available on the market, met our criteria for quality and safety.
  Other Names: Nusantara Honey
  Arms: Treatment Group (Standard Dressing and Honey)
Other: PHMB Solution — PHMB is an antimicrobial polymer that is effective against intracellular and biofilm forms of S. aureus. PHMB is quite effective in the treatment of wounds in deep neck abscesses.
  Other Names: Prontosan

SUMMARY:
This study investigates the effectiveness of honey as a treatment for deep neck space abscesses, comparing it to standard wound care methods. Conducted as a randomized clinical trial, it aims to determine whether honey can offer a viable alternative or improvement in managing this condition. The research assesses outcomes related to healing, infection control, and overall patient recovery.

DETAILED DESCRIPTION:
Deep neck abscess is one of the diseases in the field of otorhinolaryngology-head and neck surgery that has high morbidity, mortality, and costs. Management of deep neck abscesses involves incision and drainage, abscess exploration, systemic administration of broad-spectrum antibiotics, management of comorbid factors, and postoperative wound care until healing. Standard dressing for wound care has been time-consuming and costly. Honey is one type of dressing modality that has been widely used in wound care for various parts of the body and diseases. Honey is expected to be a more cost-efficient treatment modality that supports accelerated wound healing, leading to better outcomes and cost savings.

The research design used is a single-blind randomized controlled trial (RCT), where researchers randomly assign one intervention to respondents to compare the effects of honey and Prontosan on the wound healing process. The population and sample of the study include all patients with deep neck abscesses treated at Dr. Sardjito General Hospital, the teaching hospital of the Faculty of Medicine Gadjah Mada University and other hospitals equipped with board-certified Otorhinolaryngologists. The participants in the control group were treated with standard dressing, while participants in the study group were treated with standard dressing along with honey dressing.

ELIGIBILITY:
Inclusion Criteria:

* Deep neck abscess patients over 18 years old with or without comorbidities except for malignant diseases

Exclusion Criteria:

* Patients who refused intervention
* Patients who underwent vacuum-assisted closure (VAC)
* Patients with incomplete medical records

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-06-19 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Wound Assessment | BWATs was measured on the first, seventh, and fourteenth days from abscess incision.
  The wound was assessed by the research assistant using the Bates-Jensen Wound Assessment Tool
Wound Measurements | The wound was measured on the first, seventh, and fourteenth days from abscess incision.
  Wound measurements included length, width, and depth in cm, with the largest width and length used for data to report wound area in cm^2. The wound depth was measured using a probe perpendicular to the wound's length and width.
Bacterial Colony | Pus aspiration was performed by the resident doctor who conducted the dressing on the first and fourteenth days from abscess incision
  Bacterial culture results and the number of bacterial colonies served as indicators of infection improvement. Swabs from the wound bed were sent to the Microbiology laboratory.
Cytokine and Growth Factor Expression | Tissue sampling was performed by the resident doctor who conducted the dressing on the first and fourteenth days from abscess incision
  Immunopathological evaluation of wound healing involved tissue samples sent to the Anatomical Pathology laboratory for analysis of IL-1, TNF-α, and VEGF expression. Tissue sampling was performed using nasopharyngeal biopsy forceps, and the preserved tissue was sent for analysis.

SECONDARY OUTCOMES:
Vital Sign Examinations | Vital Signs were performed everyday throughout patient's admission in the wards.
  Vital signs consist of blood pressure (mmHg), heart rate per minute, respiration rate per minute, temperature (°C), and saturation (%) which are useful for monitoring patients in this study.
Blood Gas Analysis | Blood gas analysis were performed throughout patient's admission in the wards.
  Blood gas analysis showed by measuring pH, pCO2 (mmHg), HCO3 (mmol/L), pO2 (mmHg), and BE (mmol/L) status.
Complete Blood Count (CBC) | CBC were performed throughout patient's admission in the wards.
  Complete blood count performed included, Hemoglobin (g/dL), RBC (10^6/uL), WBC (10^3/uL), Platelet (10^3/uL), and blood type.
Liver Function Tests | Liver function tests were performed throughout patient's admission in the wards.
  Liver function tests typically include SGOT (U/L), SGPT (U/L), bilirubin serum (mg/dL), INR (international normalized ratio), prothrombin time (PT) and activated partial thromboplastine time (APTT) in second.
Kidney Function Tests | Kidney function tests were performed throughout patient's admission in the wards.
  Kidney function test such as albumin (g/dL), BUN (mg/dl), creatinine serum (mg/dL), uric acid (mg/dL) and electrolytes (mmol/L): sodium, potassium, chloride .
Blood Glucose Test | Blood glucose test was performed throughout patient's admission in the wards.
  A blood glucose test measure the amount of glucose in patient blood to hel diagnose or monitor diabetes either as a comorbidity or not ny doing a finger-picker test or a blood draw from patient vein

CONTACTS AND LOCATIONS:
Overall Officials: Dian Paramita Wulandari, Principal Investigator — Universitas Gadjah Mada - Dr. Sardjito General Hospital
Locations (1):
- Dr. Sardjito General Hospital, Yogyakarta, D.I Yogyakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wulandari DP, Subronto YW, Surono A. Honey as a Wound Care Modality in Treating Deep Neck Space Abscesses: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Aug 14;14:e75475. doi: 10.2196/75475. PMID 40810438